CLINICAL TRIAL: NCT03497104
Title: The Markers and Paracetamol Poisoning Study 2 - Early Diagnosis of Drug-induced Liver Injury Using Point of Care Detection of microRNA
Brief Title: The Markers and Paracetamol Poisoning Study 2
Acronym: MAPP2
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 244423
Record Dates: First submitted 2018-04-05; First posted 2018-04-13 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2022-09

CONDITIONS: Paracetamol Overdose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surplus blood tests — Surplus blood donation

SUMMARY:
Paracetamol overdose is one of the most common medical emergencies. Annually in the UK, 100,000 people seek medical attention and 50,000 need hospital admission. Treatment is with the antidote acetylcysteine (NAC), which is effective but takes 21 hours to administer intravenously and frequently produces adverse reactions.

Current tools that are used to decide who needs treatment are inadequate. this trial team have identified and validated new blood tests that accurately identify those patients at risk of liver injury by quantifying the fundamental in vivo toxicity mechanisms.

This study aim to gain further samples in order to develop a new point-of-care test specifically for the detection of liver damage.

DETAILED DESCRIPTION:
Paracetamol overdose is one of the most common medical emergencies. Annually in the UK, 100,000 people seek medical attention and 50,000 need hospital admission. Treatment is with the antidote acetylcysteine (NAC), which is effective but takes 21 hours to administer intravenously and frequently produces adverse reactions. Paracetamol is the commonest cause of acute liver failure and directly kills around 200 people/year in the UK. Management of paracetamol overdose is estimated to cost around £48 million/year to the NHS.

Current tools that are used to decide who needs treatment are inadequate. This trial team have identified and validated new blood tests that accurately identify those patients at risk of liver injury by quantifying the fundamental in vivo toxicity mechanisms. Over the last 4 years the team have published data in leading journals such as The Lancet, Lancet Gastroenterology (the MAPP Trial), Hepatology and Clinical Pharmacology & Therapeutics. The current gold standard marker, serum Alanine Aminotransferase Test (ALT) activity, lacks both sensitivity and specificity for early liver injury. This has resulted in being able to qualify 3 new liver biomarkers in over 1,200 patients (microRNA-122 (miR-122), High Mobility Group Box protein 1 (HMGB1) and keratin-18 (K18)) and demonstrated they predict liver injury at first presentation to hospital with high accuracy at a time when ALT is still normal.

This project develops a new point-of-care (POC) test for circulating microRNA specifically for the detection of liver damage after paracetamol overdose. The team have developed the microRNA biomarker (miR-122) to the point where it has received formal regulatory support from the USA Food and Drug Administration (FDA) and the European Medicines Agency (EMA). The proposed assay has backing from worldwide clinical opinion leaders and pharma partners such as AstraZeneca, GSK and Novartis. The engineering solution for POC microRNA detection is underpinned by robust pilot data and field-leading expertise. The current assay for miR-122 is PCR following extensive sample preparation which is too slow for acute clinical decision making and for dose-escalation decisions. To address this key roadblock (as identified by the FDA) the team will use electrochemical impedance spectroscopy (EIS). the trial team have over 10 years of experience in EIS-based POC test development. Pilot data demonstrate that EIS can detect miR-122 spiked into buffer and distinguish patients with DILI (high miR-122) from healthy subjects (low miR-122).

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 years and over.
2. Hospital attendance with paracetamol overdose alone or as part of a mixed overdose
3. Patient is able to give informed consent

Exclusion Criteria:

1. Patient detained under the Mental Health Act
2. Inability to provide informed consent
3. Unreliable history of overdose
4. Prisoners

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to Emergency Department or Acute Medical Unit with paracetamol overdose
Sampling Method: Non-Probability Sample
Enrollment: 464 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
To establish a biobank of human serum samples from patients with paracetamol overdose to develop and test the performance of our POC Test | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: James Dear, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.emergeresearch.org/